CLINICAL TRIAL: NCT06029972
Title: A Phase 2, Double-Blinded, Randomized, Placebo-Controlled, Dose-Ranging Study Evaluating the Efficacy and Safety of GS-5290 in Participants With Moderately to Severely Active Ulcerative Colitis
Brief Title: Study of Tilpisertib Fosmecarbil in Participants With Moderately to Severely Active Ulcerative Colitis
Acronym: PALEKONA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-457-6411; 2022-501119-14 (Other: European Medicines Agency); jRCT2031230403 (Other: Japan Registry of Clinical Trials)
Record Dates: First submitted 2023-09-01; First posted 2023-09-08 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Tilpisertib Fosmecarbil Dose A (Experimental): Blinded Treatment Phase:
  Participants will receive tilpisertib fosmecarbil Dose A for up to 12 weeks. An efficacy assessment will be performed at Week 12.
  • Participants who achieve clinical response will receive tilpisertib fosmecarbil Dose B for up to Week 52.
  Non-responder Treatment Phase:
  • Participants who do not achieve clinical response at Week 12 will discontinue the Blinded Treatment Phase and have the option to enter into the Non-responder Treatment Phase. Participants will receive tilpisertib fosmecarbil Dose A for another 12 weeks. An efficacy assessment will be performed at Week 12 of the Non-responder Treatment Phase. Participants who achieved clinical response will receive tilpisertib fosmecarbil Dose B for up to Week 52. Participants who do not achieve clinical response at Non-responder Treatment Phase Week 12 will discontinue study drug.
  Interventions: Drug: Tilpisertib Fosmecarbil
- Tilpisertib Fosmecarbil Dose B (Experimental): Blinded Treatment Phase:
  Participants will receive tilpisertib fosmecarbil Dose B for up to 12 weeks. An efficacy assessment will be performed at Week 12.
  • Participants who achieve clinical response will receive tilpisertib fosmecarbil Dose B for up to Week 52.
  Non-responder Treatment Phase:
  • Participants who do not achieve clinical response at Week 12 will discontinue the Blinded Treatment Phase and have the option to enter into the Non-responder Treatment Phase. Participants will receive tilpisertib fosmecarbil Dose B for another 12 weeks. An efficacy assessment will be performed at Week 12 of the Non-responder Treatment Phase. Participants who achieved clinical response will receive tilpisertib fosmecarbil Dose B for up to Week 52. Participants who do not achieve clinical response at Non-responder Treatment Phase Week 12 will discontinue study drug.
  Interventions: Drug: Tilpisertib Fosmecarbil
- Tilpisertib Fosmecarbil Dose C (Experimental): Blinded Treatment Phase:
  Participants will receive tilpisertib fosmecarbil Dose C for up to 12 weeks. An efficacy assessment will be performed at Week 12.
  • Participants who achieve clinical response will receive tilpisertib fosmecarbil Dose C for up to Week 52.
  Non-responder Treatment Phase:
  • Participants who do not achieve clinical response at Week 12 will discontinue the Blinded Treatment Phase and have the option to enter into the Non-responder Treatment Phase. Participants will receive tilpisertib fosmecarbil Dose B for another 12 weeks. An efficacy assessment will be performed at Week 12 of the Non-responder Treatment Phase. Participants who achieved clinical response will receive tilpisertib fosmecarbil Dose B for up to Week 52. Participants who do not achieve clinical response at Non-responder Treatment Phase Week 12 will discontinue study drug.
  Interventions: Drug: Tilpisertib Fosmecarbil
- Tilpisertib Fosmecarbil Placebo (Placebo Comparator): Blinded Treatment Phase:
  Participants will receive tilpisertib fosmecarbil placebo for up to 12 weeks. An efficacy assessment will be performed at Week 12.
  • Participants who achieve clinical response will receive tilpisertib fosmecarbil Dose C for up to Week 52.
  Non-responder Treatment Phase:
  • Participants who do not achieve clinical response at Week 12 will discontinue the Blinded Treatment Phase and have the option to enter into the Non-responder Treatment Phase. Participants will receive tilpisertib fosmecarbil Dose A for another 12 weeks. An efficacy assessment will be performed at Week 12 of the Non-responder Treatment Phase. Participants who achieved Clinical Response will receive tilpisertib fosmecarbil Dose B for up to Week 52. Participants who do not achieve Clinical Response at Non-responder Treatment Phase Week 12 will discontinue study drug.
  Interventions: Drug: Tilpisertib Fosmecarbil; Drug: Placebo

INTERVENTIONS:
Drug: Tilpisertib Fosmecarbil — Tablets administered orally
  Other Names: GS-5290
Drug: Placebo — Tablets administered orally
  Arms: Tilpisertib Fosmecarbil Placebo

SUMMARY:
The goal of this study is to learn if tilpisertib fosmecarbil (formerly known as GS-5290) is effective and safe in treating participants with moderate to severe ulcerative colitis. The study will compare participants in different treatment groups treated with tilpisertib fosmecarbil with participants treated with placebo.

The primary objective of this study is to demonstrate the efficacy of tilpisertib fosmecarbil, compared to placebo control, in achieving Clinical Response at Week 12.

ELIGIBILITY:
Key Inclusion Criteria:

* Individuals assigned male at birth, or nonpregnant, nonlactating individuals assigned female at birth, 18 to 75 years of age based on the date of the screening visit.
* Ulcerative colitis (UC) of at least 90-day duration before randomization confirmed by endoscopy and histology at any time in the past AND a minimum disease extent of 15 cm from the anal verge. Documentation of endoscopy and histology consistent with the diagnosis of UC must be available in the source documents prior to the initiation of screening.
* Moderately to severely active UC as determined during screening with a modified Mayo Clinic Score based on the sum of Stool Frequency, Rectal Bleeding, and Endoscopic Finding of 5 to 9 points and an endoscopic subscore of 2 to 3 (determined by central reader).
* Previous treatment history of approved UC therapy with at least one advanced therapy mechanisms of action but failure (ie, loss of response or lack of response) of no more than 3 different advanced therapy mechanisms of action.
* A surveillance colonoscopy for dysplasia is required prior to randomization if indicated by regional guidelines for individuals with UC.

Key Exclusion Criteria:

* Current diagnosis of Crohn's Disease (CD) or diagnosis of indeterminate colitis due to an enteric pathogen, lymphocytic or collagenous colitis.
* Individuals with disease limited to the rectum (ulcerative proctitis) during screening endoscopy.
* Requirement for ongoing therapy with or prior use of any prohibited medications.
* Active clinically significant infection, or any infection requiring hospitalization or treatment with intravenous anti-infectives within 8 weeks.

of randomization; or any infection requiring oral anti-infective therapy within 6 weeks of randomization.

* History of opportunistic infection.
* Current diagnosis of acute severe colitis, fulminant colitis, or toxic megacolon.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2023-12-05 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2028-02 (Estimated)

PRIMARY OUTCOMES:
Proportion of Participants Achieving Clinical Response Per Modified Mayo Clinic Score at Week 12 | Week 12
  Clinical Response is defined as a decrease from baseline of ≥ 2 points and at least 30% in 3 components of the modified Mayo Clinic Score, Stool Frequency, Rectal Bleeding, and Endoscopic Findings, in addition to a ≥ 1 point decrease from baseline in the Rectal Bleeding subscore or Rectal Bleeding subscore of ≤ 1. The modified Mayo Clinic Score is a scoring system for assessment of UC activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), and stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal). Total score for modified Mayo Clinic Score ranges from 0 to 9 (sum of all subscores), with higher scores indicating higher disease activity.

SECONDARY OUTCOMES:
Proportion of Participants Achieving Clinical Remission Per Modified Mayo Clinic Score at Week 12 | Week 12
  Clinical Remission is defined as a Stool Frequency subscore ≤ 1 and not greater than baseline, Rectal Bleeding subscore of 0, and Endoscopic Findings subscore ≤ 1 at Week 12. The modified Mayo Clinic Score is a scoring system for assessment of UC activity and is composed of subscores from endoscopy (range: 0 to 3, where 0 = normal or inactive disease and 3 = severe disease [spontaneous bleeding, ulceration]), rectal bleeding (range: 0 to 3, where 0 = no blood seen and 3 = blood alone passes), stool frequency (range: 0 to 3, where 0 = normal number of stools and 3 = at least 5 or more stools more than normal). Total score for modified Mayo Clinic Score ranges from 0 to 9 (sum of all subscores), with higher scores indicating higher disease activity.
Proportion of Participants Achieving Endoscopic Response at Week 12 | Week 12
  Endoscopic Response is defined as an Endoscopic Findings subscore ≤ 1 at Week 12. Endoscopic subscore is a part of the modified Mayo Clinic Score which is a scoring system for assessment of UC activity. Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern), 2 = moderate disease (marked erythema, lack of vascular pattern, friability, erosions), and 3 = severe disease (spontaneous bleeding, ulceration). Higher scores indicate higher disease activity.
Proportion of Participants Achieving Histologic Endoscopic Mucosal Improvement at Week 12 | Week 12
  Histologic Endoscopic Mucosal Improvement is defined as an Endoscopic Findings subscore ≤ 1 and Geboes score ≤ 3.1 (indicating neutrophil infiltration in < 5% of crypts, no crypt destruction and no erosions, ulcerations, or granulation tissue). Endoscopic subscore is a part of the modified Mayo Clinic Score which is a scoring system for assessment of UC activity. Endoscopic subscore range: 0 to 3, where 0 = normal or inactive disease, 1 = mild disease (erythema, decreased vascular pattern), 2 = moderate disease (marked erythema, lack of vascular pattern, friability, erosions), and 3 = severe disease (spontaneous bleeding, ulceration). Geboes histologic remission is assessed using the Geboes histologic scores to identify histologic changes in ulcerative colitis. Possible scores are graded as Grade 0 to Grade 5, with higher grade representing higher levels of disease activity.
Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | First dose date up to Week 52 (responders) or Week 64 (non-responders) plus 30 days
Percentage of Participants Experiencing Clinically Significant Laboratory Abnormalities | First dose date up to Week 52 (responders) or Week 64 (non-responders) plus 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (129):
- United States (53):
  - GI Alliance, Sun City, Arizona
  - GastroSb Weight Loss Clinic, Chula Vista, California
  - Southern California Research Centers, Coronado, California
  - VVCRD Research, Garden Grove, California
  - UC San Diego Health System, La Jolla, California
  - Gastro Care Institute, Lancaster, California
  - Om Research LLC, Lancaster, California
  - United Medical Doctors, Murrieta, California
  - University of California, Davis, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Amicis Research Center, Valencia, California
  - Luna Research, Coral Gables, Florida
  - University of Florida, Gainesville, Florida
  - The Medici Medical Research, Hollywood, Florida
  - Encore Medical Research, LLC, Hollywood, Florida
  - Clinical Research of Osceola, Kissimmee, Florida
  - Florida Research Institute, Largo, Florida
  - Wellness Research Center, Miami, Florida
  - IMIC Inc, Miami, Florida
  - Reserka LLC, Miami, Florida
  - GI PROS Research, Naples, Florida
  - Clinical One Research, Orlando, Florida
  - Digestive and Liver Center of Florida, LLC, Orlando, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Gastroenterology Associates of Florida - GI Alliance, Wellington, Florida
  - Atlanta Center For Gastroenterology P.C., Decatur, Georgia
  - Corewell Health, Grand Rapids, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Gastroenterology Associates of North Mississippi, Oxford, Mississippi
  - Digestive Health Specialists, Tupelo, Mississippi
  - St. Charles Clinical Research, St Louis, Missouri
  - Ellipsis Research Group, Brooklyn, New York
  - NYU Langone Long Island Clinical Research Associates, Great Neck, New York
  - Gastroenterology & Hepatology Specialists Inc, Canton, Ohio
  - Ohio Gastroenterology & Liver Institute, Cincinnati, Ohio
  - The Ohio State University Wexner Medical Centre, Columbus, Ohio
  - Dayton Gastroenterology, LLC, Dayton, Ohio
  - Great Lakes Gastroenterology Research, LLC, Mentor, Ohio
  - Hightower Clinical, Oklahoma City, Oklahoma
  - Skyline Gastroenterology of West Tennessee, Jackson, Tennessee
  - Gastroenterology Research of Hill Country, Boerne, Texas
  - Gastroenterology Research of America, El Paso, Texas
  - DHAT Research Institute, Garland, Texas
  - Southwest Clinical Trials, Houston, Texas
  - GI Alliance, Lubbock, Texas
  - GI Associates and Endoscopy Center - GI Alliance, Mansfield, Texas
  - Clinical Associates in Research Therapeutics of America, San Antonio, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Tyler Research Institute, LLC, Tyler, Texas
  - Gastroenterology Associates of Tidewater, Chesapeake, Virginia
  - Emeritas Group Research, Lansdowne Town Center, Virginia
  - Gastroenterology Consultants of Southwest Virginia, Roanoke, Virginia
  - Swedish Medical Center, Seattle, Washington
- Australia (9):
  - Sunshine Coast University Hospital, Birtinya, Queensland
  - Mater Adult Hospital, South Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Queen Elizabeth Hospital, Woodville, South Australia
  - Monash Medical Centre, Clayton, Victoria
  - Northern Health, Epping, Victoria
  - Footscray Hospital, Footscray, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Austria (4):
  - Medical University of Innsbruck, Innsbruck
  - University of Salzburg, Universitätsklinik für Innere Medizin III, Salzburg
  - Universitätsklinikum St. Pölten, Sankt Pölten
  - Medical University Vienna, Department of Internal Medicine III, Division Gastroenterology and Hepatology, Vienna
- Universitaire Ziekenhuis Leuven, Leuven, Belgium
- Canada (4):
  - London Health Sciences Centre-University Hospital, London
  - Physician's Clinical Research, Inc. (PCRI), Toronto
  - Mount Sinai Hospital, Toronto
  - TDDA Speciality Research, Vaughan
- France (8):
  - Centre Hospitalier Universitaire Grenoble, Grenoble
  - Hôpital Claude Huriez, Little Cedex
  - Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire de Nantes, Nantes
  - Institut des MICI, Neuilly-sur-Seine
  - CHU de Saint Etienne - Hopital Nord, Saint-Etienne
  - Hopital Rangueil, Toulouse
  - CHRU Nancy, Vandœuvre-lès-Nancy
- Germany (5):
  - Charite Universitaetsmedizin Berlin Campus CVK, Department of Hepatology and Gastroenterology, Berlin
  - Medizinische Hochschule Hannover, Hanover
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Eugastro Gmbh, Liepzig
  - Universitaetsklinikum Ulm Klinik fur Innere Medizin I CED Studien Ambulanz, Ulm
- Hungary (2):
  - Tolna Megye Balassa Janos Korhaz, Beri Balogh
  - Szent Janos Korhaz es Eszak-budai Egyesitett Korhazak, Budapest
- Italy (5):
  - AZIENDA UNICA OSPEDALIERO-UNIVERSITARIA"RENATO DULBECCO" - AOU"Mater Domini", Catanzaro
  - IRCCS Istituto Clinico Humanitas, Milan
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Istituto Clinico Humanitas, Rozzano
  - Azienda Sanitaria Universitaria Friuli Centrale, Udine
- Japan (12):
  - Hyogo Medical University Hospital, Hyōgo
  - Fukuoka University Hospital, Jonan-ku
  - The Jikei University Hospital, Minatoku
  - Kitasato University Kitasato Institute Hospital, Minatoku
  - Kyorin University Hospital, Mitaka-shi
  - Nagasaki University Hospital, Nagasaki
  - Ishida Clinic of IBD and Gastroenterology, Ōita
  - Saga University Hospital, Sagaken
  - Kitasato University Hospital, Sagamihara
  - Sapporo Medical University Hospital, Sapporo
  - Ginza Central Clinic, Tokyo
  - Institute of Science Tokyo Hospital, Toukiyouto
- Poland (11):
  - Economicus Sp. z o.o., Niepubliczny Zakład Opieki Zdrowotnej (NZOZ) ALL-MEDICUS, Katowice
  - Gabinet Endoskopii Przewodu Pokarmowego, Krakow
  - Medrise Sp. z o.o. Centrum Badań Klinicznych, Lublin
  - SOLUMED Centrum Medyczne, Poznan
  - Kliniczny Szpital Wojewódzki Nr 2 im. Sw. Jadwigi Królowej w Rzeszowie, Rzeszów
  - Specjalistyczna Praktyka Lekarska Leszek Bryniarski, Sopot
  - GASTROMED Kopon, Zmudzinski i wspolnicy Sp. J. Specialized Center of Gastroenterology and Endoscopy, Torun
  - Medical Network Sp. z o.o. WIP Warsaw IBD Point Profesor Kierkus, Warsaw
  - Nzoz Vivamed, Warsaw
  - Specjalistyczne Gabinety Lekarskie Body Clinic, Warsaw
  - Centrum Medyczne Oporow, Wroclaw
- South Korea (9):
  - Yonsei University Severance Hospital, Seodaemun-Gu, VIC
  - Inje University, Busan
  - Yeungnam University Hospital, Daegu
  - Kyungpook National University Hospital, Junggu
  - Kyung Hee University Medical Center, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Hanyang University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
- Intesto, Gastroenterologische Praxis Crohn-Colitis-Zentrum, Bern, Switzerland
- United Kingdom (5):
  - Fairfield General Hospital, Bury
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - Barts Health NHS Trust, London
  - Norfolk and Norwich University Hospital Nhs Foundation Trust, Norwich
  - University Hospital Southampton Nhs Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.gileadclinicaltrials.com/study?nctid=NCT06029972